CLINICAL TRIAL: NCT00002356
Title: An Open-Label Study of the Safety and Efficacy of Intravitreal ISIS 2922 in Acquired Immune Deficiency Syndrome (AIDS) Patients With Cytomegalovirus Retinitis (NOTE: Restricted to Patients Who Rollover From Another Controlled ISIS 2922 Trial)
Brief Title: The Safety and Effectiveness of ISIS 2922 in Patients With AIDS Who Have Cytomegalovirus (CMV) of the Eyes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 251C; ISIS 2922-CS7
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Antiviral Agents; Cytomegalovirus Retinitis
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — fomivirsen

INTERVENTIONS:
Drug: Fomivirsen sodium

SUMMARY:
To evaluate the efficacy and safety of ISIS 2922 in AIDS patients with Cytomegalovirus ( CMV ) retinitis who are unresponsive or intolerant to ganciclovir and/or foscarnet but are otherwise ineligible for ISIS Pharmaceuticals' controlled trials OR who have failed ISIS 2922 therapy on another controlled clinical trial.

PER 2/8/96 AMENDMENT: Patients must rollover from another ISIS 2922 controlled trial.

DETAILED DESCRIPTION:
Patients receive intravitreal injections of ISIS 2922 at doses of either 150 or 300 mcg, depending on CMV retinitis location and extent of retinal involvement. There is a 3-week Induction period followed by at least 18 weeks of Maintenance. Induction is given on days 1, 8, and 15, and Maintenance doses are given every 14 days, beginning on day 29.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS.
* CMV retinitis in one or both eyes that was previously treated but is presently uncontrolled.
* Intolerance or resistance to other therapies.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Eligibility to participate in a controlled clinical trial of ISIS 2922.
* External ocular infection in eye to be treated.
* Other herpetic infections of the retina, toxoplasma retinochoroiditis, or other diseases of the fundus in eye to be treated.
* Ocular condition that would obstruct visualization of the posterior ocular structures in eye to be treated.
* Retinal detachment in eye to be treated.
* Known or suspected allergy to phosphorothioate oligonucleotides.
* Silicone oil in eye to be treated.
* Syphilis.
* Clinical evidence of retinal pigment epithelial stippling.
* Pseudoretinitis pigmentosa.

Concurrent Medication:

Excluded:

* Foscarnet.
* Mellaril, Stelazine, Thorazine, and Clofazimine.
* Ethambutol / fluconazole combination.
* Other investigational drugs for CMV retinitis.

Patients with the following prior conditions are excluded:

* History of surgery to correct retinal detachment in eye to be treated.
* History of ganciclovir implant for treatment of CMV retinitis.
* History of intolerance to ISIS 2922.
* History of syphilis.

Required:

* Prior CMV retinitis therapy with ganciclovir, foscarnet, or ISIS 2922.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - UCI College of Medicine, Irvine, California
  - Retina - Vitreous Associates Med Group, Los Angeles, California
  - Community Eye Med Group, Pasadena, California
  - San Diego Naval Hosp, San Diego, California
  - Univ of California San Francisco / SF Gen Hosp, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Dr Alan Palestine, Washington D.C., District of Columbia
  - Dr Julio Perez, Fort Lauderdale, Florida
  - Bascon Palmer Eye Institute, Miami, Florida
  - Emory Univ School of Medicine / Emory Eye Ctr, Atlanta, Georgia
  - Georgia Retina, Atlanta, Georgia
  - Univ of Illinois, Chicago, Illinois
  - Indiana Univ Med Ctr, Indianapolis, Indiana
  - Tulane Univ, New Orleans, Louisiana
  - Vitreo - Retinal Consultants, New York, New York
  - Charlotte Eye Ear Nose & Throat Association, Charlotte, North Carolina
  - Duke Univ, Durham, North Carolina
  - Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Graduate Hosp, Philadelphia, Pennsylvania
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia
  - Novum Inc, Seattle, Washington